CLINICAL TRIAL: NCT00854074
Title: Neurostimulation for the Treatment of Post-Operative Ileus
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn: study halted prematurely, prior to enrollment of first participant
Sponsor: ElectroCore INC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IL - 01
Record Dates: First submitted 2009-02-26; First posted 2009-03-02 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Ileus
Keywords: Post-operative Paralytic Ileus; Neuromodulation; Neurostimulation; Extended loss of functional bowel motility
MeSH Terms: conditions — Ileus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (No Intervention): Subject will be observed until recovery of normal GI function
- 1 (Experimental): Spinal neurostimulation
  Interventions: Device: ElectroCore RMS-1100 Resolution Motility System™

INTERVENTIONS:
Device: ElectroCore RMS-1100 Resolution Motility System™ — An electrical neurostimulation signal will be applied to the spine
  Arms: 1

SUMMARY:
The primary goal of this study is to validate the design of the ElectroCore RMS-1100 Resolution Motility System™ and the ability to safely place a stimulation electrode in the epidural space of the spine in a post-operative subject, and to evaluate the subject's ability to tolerate stimulation for up to 48 hours. The secondary goal is to confirm that the electrical signal being delivered via this electrode shows evidence of effectiveness in improving the functional GI motility in subjects experiencing post-operative paralytic ileus

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effects of neurostimulation in the epidural space in the spine on the activity of the enteric nervous system (ENS).

ElectroCore has successfully studied POI in an animal model and believes that temporary neurostimulation of the spine may be useful in re-starting the ENS in humans, resulting in the resumption of coherent GI motility in the gut and normal bowel function in a shorter period of time than currently occurs. Electrical pulses will be used to modulate the signals that may be preventing a return to normal GI activity. This device and procedure used in this study are similar to the system and procedure used to implant the temporary trial stimulator used evaluate the effectiveness of spine pain stimulation prior to implantation of the permanent device.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, Age >18 years, < 65 years
* Partial small or large bowel open resection with primary anastomosis
* 120 hours post-operative with no signs of functional bowel activity
* Able to give Informed Consent
* By Post-Op Day 5, patient care has involved at least 3 of the following conservative therapies to minimize long term POI:

  i. post-operative, patient controlled opioid analgesia ii. removal of intra-operative nasogastric tube at time of surgery or on post-operative day 1 iii. advancement of liquid diet iv. advancement of solid food v. ambulation vi. use of chewing gum

Exclusion Criteria:

* Pregnant
* Undergoing surgery for repair of penetrating trauma injury, gangrene or ischemic bowel
* Evidence of anastomotic leak, abdominal infection, sepsis, bowel perforation, mechanical small bowel obstruction or metabolic derangement (e.g., low potassium/magnesium)
* Presence of existing implanted or external stimulator for pain or other indications (including pacemaker)
* Operative blood lost of > 500 cc
* Significant scarring of the skin along the lower thoracic/lumbar spine or deformation of thoracic spinal canal from congenital, developmental or traumatic causes, or previous extensive spinal thoracic surgery other than diskectomy
* Received a lumbar or thoracic epidural block placed immediately prior to surgery
* Body Mass Index > 35
* Unstable cardiac status
* Severe hypertension
* American Society of Anesthesiologists (ASA) Score greater than/equal to 3
* On anti-coagulation therapy (other than aspirin) or has an underlying bleeding disorder
* Active or suspected pelvic infection
* Unable to communicate perception of the stimulation
* Significant surgical complications where in the view of the physician, participation in the study could further complicate subject care (i.e. infection at surgical site, deep venous thrombosis, respiratory complications, etc)
* Treatment with Entereg (alvimopam) during post-operative period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-07; Primary Completion 2009-12 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
To validate the design of ElectroCore Resolution Motility System™ , to safely place a stimulation electrode in the epidural space of the spine in a post-operative subject, and to evaluate the subject's ability to tolerate stimulation for up to 48 hours | 30 days

SECONDARY OUTCOMES:
To confirm that the electrical signal being delivered via this electrode shows evidence of effectiveness in improving the functional motility in subjects experiencing post-operative paralytic ileus. | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Michael Erdeck, MD, Principal Investigator — Johns Hopkins Medical Center; David Walega, MD, Principal Investigator — Northwestern University Medical Center; Robert Frye, MD, Principal Investigator — Pennsylvania Hospital
Locations (3):
- United States (3):
  - Northwestern, Chicago, Illinois
  - Johns Hopkins Medical Center, Baltimore, Maryland
  - Pennsylvania Hospital, Philadelphia, Pennsylvania